CLINICAL TRIAL: NCT04101214
Title: Effects of Dry Needling on Function, Muscle Tone and Quality of Life in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Collaborators: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNHS_Parkinson
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease
Keywords: Dry needling; Parkinson Disease; myofascial trigger point
MeSH Terms: conditions — Parkinson Disease | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking is with sham dry needling, simulating to insert the needle, so no real masking 100%
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): One session of dry needling technique will be applied by a physiotherapist specialized in the technique. Dry needling technique will be performed in the muscle of the lower limb whose MMAS score is >1 by locating a sensitive point within a taut band. After that, a thin needle (0,32x40mm) is introduced directly into those muscle that present spasticity, decide by the clinician expert.
  Interventions: Other: Dry needling
- Sham Dry needling (Sham Comparator): A physiotherapist specialized in dry needling technique will use a sham needle in order to simulate the active intervention. Sham acupuncture uses non-penetrating needles.The palpation and evaluation of the spastic muscle will be exactly the same that in the active group.
  Interventions: Other: Sham dry Needling

INTERVENTIONS:
Other: Dry needling — Dry needling into spastic muscle
  Other Names: DNHS technique
  Arms: Dry needling
Other: Sham dry Needling — Sham dry needling into spastic muscle
  Arms: Sham Dry needling

SUMMARY:
Hypothesis: Dry needling in lower limbs produces a change in function (assessed by the 6 minute walk test, timed up and go, 10 meter walk test and unified scale for Parkinson's disease) and muscle tone (assessed by tonometry and the modified of Modified Ashworth scale(MMAS)) in patients with Parkinson's disease.

The main objective of this study is to analyze the effect of dry needling on function and muscle tone in subjects with Parkinson disease.

The secondary objective is to analyze the longterm effects of dry needling on function and muscle tone in subjects with Parkinson disease.

DETAILED DESCRIPTION:
Methods:

It is a double-blinded randomized clinical trial where subjects are patients from Zaragoza and have been diagnosed with Parkinson´disease by a neurologist.

Inclusion criteria:

* Patients diagnosed with Parkinson by a neurologist.
* Age: 50 - 90 years.
* Presence of Hypertonia according to: MMAS score > 1 during movement of ankle dorsiflexion or knee flexion and extension.

Exclusion criteria:

* Degenerative diseases that may affect the results.
* Presence of fixed contractures.
* Fear of needles.
* No tolerance to pain caused by dry needling
* No commitment to continuity.
* Attrition criteria

Attrition criteria:

* Adverse effects relate to the DNHS technique.
* Subject Uncooperative that prevents proper protocol execution performance -Voluntary decision of the patient.

Intervention:

There will be an intervention group (dry needling into the muscles of the lower limbs that present tone dysfunction according to an expert clinician) and a control group (sham dry needling). The intervention will be a unique session.

Dry needling technique will be performed by locating the taut band and the Myofascial Trigger Point by an expert clinician. After that, a thin needle (0,32x40mm) is introduced directly into a Myofascial Trigger Point with the aims to generate a "local twitch response" that are involuntary contractions of the muscle fibers. This puncture may reproduce patient's symptoms, and causes muscle relaxation to achieve at the same time the relief of muscle tension and pain and also to recover the metabolism of the muscle.

Assessment:

Outcome measures will include tone muscle measured by tonometry and the MMAS and functional clinical scales including: 6 minute walk test, timed up and go, 10 meter walk test and Unified Parkinson's Disease Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Parkinson by a neurologist
* Age: 50 - 90 years
* Presence of Hypertonia according to: MMAS score > 1 during movement of ankle dorsiflexion or knee flexion and extension

Exclusion Criteria:

* Degenerative diseases that may affect the results.
* Presence of fixed contractures.
* Fear of needles
* No tolerance to pain caused by dry needling
* No commitment to continuity

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
6 minute walk test | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). Change between baseline (immediately before intervention) and follow-up (at 1 week after intervention)
  It measures the maximum distance that the subject is able to travel in 6 minutes. It allows to obtain the speed of walking.
Timed up and go test | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). Change between baseline (immediately before intervention) and follow-up (at 1 week after intervention)
  It measures patient mobility. The patient should get up from a chair with armrests, walk three meters, turn on himself, step back three meters and sit back down. If the patient takes less than 10s, it is considered normal mobility and more than 20s reduced mobility
10 meter walk test | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). Change between baseline (immediately before intervention) and follow-up (at 1 week after intervention)
  It used to assess walking speed in meters/second (m/s) over a short distance

SECONDARY OUTCOMES:
Modified Modified Ashworth score | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). Change between baseline (immediately before intervention) and follow-up (at 1 week after intervention)
  Scale measuring Spasticity/Hypertonia. This scale ranges from 0 to 4 points for each muscle assessed, where 0 is no hypertonia/spasticity and 4 is the highest hypertonia/spasticity.
Tonometry (measurement of muscle tone with a device) | Change between baseline (immediately before intervention) and post intervention (immediately after intervention). Change between baseline (immediately before intervention) and follow-up (at 1 week after intervention)
  Muscle stiffness or muscle tone (Quadriceps, Hamstring, soleus and gastrocnemius). This device register different parameters like frequency, oscillation, etc that are related to tone, and start from 0 to an undefined number (depending on every muscle). It is a quantitative measurement.
  It is a quantitative measurement.
Unified Parkinson's Disease Rating Scale | Change between baseline (immediately before intervention) and follow-up at 1 week after intervention
  It measures the motor and cognitive function, the activities of daily life, as well as the possible complications that can alter the patient's life. The score ranges from 0 to 199, where 199 represents total disability and 0 no disability

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Bravo, Phd, Study Director — University of Castilla-La Mancha
Locations (1):
- Asociación de Parkinson de Aragón, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No